CLINICAL TRIAL: NCT00245583
Title: Topiramate in the Treatment of Pathological Gambling: A Randomized, Double-Blind, Placebo-Controlled, Flexible-Dose Study
Brief Title: Topiramate in the Treatment of Pathological Gambling
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: low enrollment
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Ortho-McNeil, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAPSS-314; GCO 04-0023PS*; NCT00277628 (obsolete NCT alias)
Record Dates: First submitted 2005-10-26; First posted 2005-10-28 (Estimated); Results first posted 2019-07-02 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-07

CONDITIONS: Pathological Gambling
Keywords: Pathological Gambling; Compulsive Gambling; Gambling; topiramate
MeSH Terms: conditions — Gambling | interventions — Topiramate

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Topiramate (Experimental): 25mg to 300mg daily dose
  Interventions: Drug: Topiramate
- Placebo (Placebo Comparator): placebo equivalent tablets
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Topiramate — minimum does of 50mg/day
  Other Names: Topamax
  Arms: Topiramate
Drug: Placebo — matching tablet
  Arms: Placebo

SUMMARY:
This study will assess the efficacy of topiramate in the treatment of pathological gambling. Pathological gambling (PG) is a debilitating disorder, generally leading to severe personal, familial, financial, social, and occupational impairments. In PG, the patient experiences a progressive inability to resist impulses to gamble, and gambling significantly disrupt the patient's functioning in the personal, familial, and/or vocational spheres. Topiramate has shown preliminary evidence of efficacy in some impulse control disorders.

DETAILED DESCRIPTION:
This is a 14-week, outpatient, multicenter, randomized, double-blind, placebo-controlled, flexible-dose study of topiramate in subjects with pathological gambling. After giving informed consent, subjects who meet all the inclusion and exclusion criteria may be enrolled. The study will consist of three phases:

* Washout/Screening Phase (up to 28 days prior to randomization or longer for those medications requiring a longer washout period;
* Double-Blind Phase (Titration: up to 6 weeks; Maintenance: 8 weeks); and
* Taper Phase (approximately 1 week).

The study medication will be titrated to 300 mg/day or the subject's maximum tolerated dose (MTD). Subjects must reach a minimum dose of 50 mg/day by Week 2. The taper phase will last approximately one week where subjects gradually reduce their medication until they are no longer taking study medication.

Patient may also give an optional blood sample for pharmacogenomic testing

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a current DSMV-IV-TRTM diagnosis of pathological gambling supported by the Structured Clinical Interview for Pathological Gambling (SCI-PG).
* Subjects must have a severity score of ³ 4 (moderately ill) on the Clinical Global Impressions Scale - Severity (CGI-S) at Visit 1A (Day -28).
* Subjects must have a severity score of ³5 on the South Oaks Gambling Screen (SOGS) at Visit 1B (Day -7).
* Subjects must have a score of ³2 for item number 1 on the Gambling Symptom Assessment Scale (G-SAS) at Visit 1B (Day -7) and Visit 2 (Day 1).
* Subjects must have a minimum score of >10 on the obsession subscale (questions 1-5) of the Pathological Gambling - Yale Brown Obsessive Compulsive Scale (PG-Y-BOC) at Visits 1B (Day -7) and 2 (Day 1).
* Subjects must score ≤15 on the Young Mania Rating Scale (YMRS) at Visits 1B (Day -7) and 2 (Day 1).
* Subjects must be between 18 and 70 years of age, inclusive.
* Subjects must provide contact information for themselves to be used by the site in case of a missed appointment.
* Subjects may be male or female and must be in generally good health as confirmed by medical history and physical examination, laboratory tests and vital signs.
* Female subjects must be:

  * postmenopausal for at least one year, or
  * surgically sterile, or
  * practicing an effective method of birth control (e.g., oral contraceptives, contraceptive injections, intrauterine device, spermicide with barrier, contraceptive patch, contraceptive vaginal ring, male partner sterilization, or abstinence and agree to continue abstinence or to use an acceptable method of contraception, as listed above, should sexual activity commence) before entry and throughout the study; have a negative urine pregnancy test at Visits 1B (Day -7) and 2 (Day 1).
* Subjects must be able to take oral medication, adhere to the medication regimens and be willing to return for regular visits.
* Subjects must be able and willing to read written instructions and complete all scales and inventories required by the protocol.
* Subjects must have signed an informed consent form indicating that they understand the purpose of and procedures required for the study and are willing to participate.

Exclusion Criteria:

* Subjects with any current Axis I psychiatric disorder as defined by DSM-IV-TRä supported by the SCID-I/P, other than pathological gambling, that in the investigator's judgment might require intervention with either pharmacological or non-pharmacological therapy over the course of the study.
* Subjects with a history of personality disorder (e.g., schizotypal or borderline) considered by the investigator to likely interfere with assessment or compliance with treatment.
* Subjects who have a current or recent (within 3 months of Visit 2, Day 1) DSM-IV-TRTM diagnosis of substance abuse or dependence, with the exception of nicotine and caffeine abuse or dependence.
* Subjects receiving formal psychotherapy for pathological gambling (with the exception of Gamblers Anonymous) within the 4 weeks prior to Visit 1B (Day -7).

Note: Formal psychotherapy is defined as behavioral therapy, cognitive therapy, cognitive-behavioral therapy, psychoanalysis, etc. for the treatment of a clinical diagnosis or for which a healthcare professional is billing for such therapy.

- Subjects who have begun to receive formal psychotherapy for a psychiatric disorder, other than pathological gambling, within 3 months prior to Visit 1B (Day -7).

Note: Subjects who have been engaged in formal psychotherapy for a condition other than pathological gambling for >3 months and plan to maintain therapy throughout the study will be considered on a case-by-case basis.

* Subjects with a score of >24 on the Montgomery-Asberg Depression Rating Scale (MADRS) at Visit 1B (Day -7) and Visit 2 (Day 1).
* Subjects who are expected to stay in a restricted environment.
* Subjects who have taken a prohibited medication described in the Concomitant Therapy section of the protocol and who have not met the washout criteria specified in Attachment 15.
* Subjects with a positive urine drug screening [benzodiazepines, phencyclidine, cocaine, amphetamines, tetrahydrocannabinol (THC), and opiates] at Visit 1B (Day -7).

Note: Subjects with a positive urine drug screen for THC may be retested in 7 days and enrolled if they a) continue to meet inclusion/exclusion criteria and b) have a negative urine drug screen upon retest.

* Subjects who are pregnant or lactating.
* Subjects who are members of the same household.
* Subjects with a history of nephrolithiasis.
* Subjects known to have clinically significant medical conditions, including but not limited to:

  1. symptomatic coronary artery disease or peripheral vascular disease;
  2. malignancy or history of malignancy within the past 5 years (except basal cell carcinoma);
  3. renal disease and/or impaired renal function as defined by subjects with an estimated creatinine clearance of £60 mL/min;
  4. diseases of the gastrointestinal system including active liver disease;
  5. subjects with AST and/or ALT >2 times the upper limit of the normal range and/or an increased serum bilirubin > 2.0 mg/dL at Visit 1B (Day -7); Note: if these values are abnormal they can be re-tested prior to enrollment. If the repeat study is within the limits of the protocol the subject may be randomized.
  6. pulmonary disorders including subjects with active tuberculosis;
  7. endocrinological disorders;
  8. neurological disorders including subjects with seizure disorders and subjects with progressive or degenerative neurological disorders (e.g., multiple sclerosis); or I. any disease or condition that compromises the function of those body systems that could result in altered absorption, excess accumulation, or impaired metabolism or excretion of topiramate.
* Subjects who have previously been treated with topiramate for any reason and discontinued treatment due to an adverse event or a hypersensitivity reaction to topiramate.
* Subjects with prior non-response to topiramate for the treatment of pathological gambling following an adequate trial.
* Subjects who in the opinion of the investigator should not be enrolled in the study because of the precautions, warnings or contraindications outlined in the topiramate investigator brochure and/or package insert.
* Employees of the investigator or study center, with direct involvement in the proposed study or other studies under the direction of that investigator or study center, as well as family members of the investigator or study center employees.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2005-10; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Hollander, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai School of Medicine, New York, New York, United States

REFERENCES:
- [Result] Berlin HA, Braun A, Simeon D, Koran LM, Potenza MN, McElroy SL, Fong T, Pallanti S, Hollander E. A double-blind, placebo-controlled trial of topiramate for pathological gambling. World J Biol Psychiatry. 2013 Mar;14(2):121-8. doi: 10.3109/15622975.2011.560964. Epub 2011 Apr 12. PMID 21486110

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited primarily through community advertisements such as newspapers and targeted advertisements in casinos. Eligible participants were enrolled between October 26, 2005 and May 23, 2008.
Pre-assignment Details: Subjects were randomized in a 1:1 ratio to topiramate or placebo treatment. Following the baseline visit, participants underwent a 6-week titration period to 300mg/day or the maximum tolerated dose, followed by an 8-week maintenance. At the conclusion of the 14-weeks, study medication was tapered over a 7-day period.
Period: Overall Study
Arm/Group | Topiramate | Placebo
Started | 20 | 22
Completed | 14 | 13
Not Completed | 6 | 9
Not completed — Lost to Follow-up | 1 | 5
Not completed — Adverse Event | 2 | 1
Not completed — Lack of Efficacy | 1 | 0
Not completed — Withdrawal by Subject | 2 | 3

BASELINE CHARACTERISTICS:
Population: Pathological Gamblers meeting criteria
Groups:
- Total: Total of all reporting groups
Arm/Group | Topiramate | Placebo | Total
Number analyzed (Participants) | 20 | 22 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.45 (10.44) | 44.91 (8.01) | 47.5 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 15 | 23
  Male | 12 | 7 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 5 | 12
  White | 11 | 16 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Smoking [Number; unit: participants]
  Smoker | 8 | 15 | 23
  Non-smoker | 12 | 7 | 19

OUTCOME MEASURES:

1. Primary Outcome: Obsession Component of the Yale-Brown Obsessive-Compulsive Scale for Pathological Gambling (PG-YBOCS)
Description: The obsessions subscale of the Yale-Brown Obsessive Compulsive Scale modified for PG (PG-YBOCS) measures the severity and change in severity of PG symptoms such as thoughts/urges and behaviors and has been shown to be reliable and valid and correlate with global severity and South Oaks Gambling Screen scores. The scale is a clinician-rated, each item rated from 0 (no symptoms) to 4 (extreme symptoms), Each component, Obsession and Compulsion, score ranges from 0-20, yielding a total possible score range from 0 to 40, with higher score indicating more symptoms.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Topiramate | Placebo
Number analyzed (Participants) | 20 | 22
score on a scale
  Obsessions | 12.65 (2.08) | 12.95 (2.24)
  Compulsions | 11.10 (23.75) | 12.27 (2.91)
  Total | 23.75 (4.80) | 25.23 (4.89)

2. Primary Outcome: Obsession Component of the Yale-Brown Obsessive-Compulsive Scale for Pathological Gambling (PG-YBOCS)
Description: as for outcome 1
Time Frame: 14 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Topiramate | Placebo
Number analyzed (Participants) | 14 | 13
score on a scale
  Obsessions | 6.17 (3.28) | 7.62 (3.66)
  Compulsions | 5.28 (4.71) | 6.92 (4.48)
  Total | 11.44 (7.81) | 14.54 (7.79)

3. Secondary Outcome: Gambling-Symptom Assessment Scale Total Score
Description: The Gambling-Symptom Assessment Scale (G-SAS) is a 12-item self-rated measure that is designed to assess gambling symptom severity and change during treatment. Each item is scored on a 4 point scale from 0-4 with 0 meaning no symptoms and 4 meaning extreme symptoms. The total score is 0 - 48, with higher score indicating more gambling problem. Scores 7 and lower are considered normal behavior, 8-20 are considered a mild gambling problem, 21-30 are considered a moderate gambling problem, 31-40 are considered a severe gambling problem and 40-48 are considered an extreme gambling problem.
Time Frame: baseline and 14 weeks
Population: those who returned for week 14 visit included in data results
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Topiramate | Placebo
Number analyzed (Participants) | 20 | 22
score on a scale
  baseline | 31.95 (7.41) | 35.73 (7.85)
  14 weeks: number analyzed (Participants) | 14 | 13
  14 weeks | 19.94 (9.18) | 23.00 (11.55)

4. Secondary Outcome: Barratt Impulsiveness Scale-11
Description: The Barratt Impulsiveness Scale (BIS-11) is a questionnaire designed to assess the personality/behavioral construct of impulsiveness, composed of 30 items describing common impulsive or non-impulsive (for reverse scored items) behaviors and preferences. Subscale attentional score 8-32, subscale motor score 11-44, subscale nonplanning score 11-44, with higher scores for each subscale indicating worse outcomes. Total score from 30-120, with higher score indicating more impulsive symptoms. Items are scored on a 4-point scale:
  Rarely/Never = 1 Occasionally = 2 Often = 3 Almost Always/Always = 4 Total scores of 72+ = high impulsiveness Total scores between 52 and 71 = within normal limits for impulsiveness Total scores lower than 52 are representative of an individual that is either extremely over-controlled or who has not honestly completed the questionnaire
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Topiramate | Placebo
Number analyzed (Participants) | 20 | 22
score on a scale
  Attentional | 18.18 (4.03) | 18.00 (4.57)
  Motor | 25.35 (3.83) | 25.27 (4.86)
  Non-planning | 30.07 (3.91) | 28.90 (5.50)
  Total | 73.59 (9.22) | 72.16 (12.50)

5. Secondary Outcome: Barratt Impulsiveness Scale-11
Description: as for outcome 4
Time Frame: week 14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Topiramate | Placebo
Number analyzed (Participants) | 14 | 13
score on a scale
  Attentional | 16.83 (4.3) | 17.41 (5.13)
  Motor | 22.32 (3.37) | 23.85 (5.05)
  Non-planning | 29.00 (4.04) | 30.38 (6.10)
  Total | 68.14 (8.30) | 71.66 (14.54)

6. Secondary Outcome: Young Mania Rating Scale (YMRS)
Description: The YMRS is an 11-item scale used to assess the severity of mania and is based on the patient's subjective report of his or her clinical condition over the previous 48 hours. Additional information is based upon clinical observations made during the course of the clinical interview. There are four items that are graded on a 0 to 8 scale (irritability, speech, thought content, and disruptive/aggressive behavior), while the remaining seven items are graded on a 0 to 4 scale. These four items are given twice the weight of the others to compensate for poor cooperation from severely ill patients. YMRS total score varies between zero and 60, with higher score indicating more symptoms. A score of <= 12 indicates remission of symptoms.
Time Frame: baseline and week 14
Population: those who returned for week 14 visit included in data results
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Topiramate | Placebo
Number analyzed (Participants) | 20 | 22
score on a scale
  Baseline | 3.85 (3.65) | 3.95 (3.84)
  14 weeks: number analyzed (Participants) | 14 | 13
  14 weeks | 2.61 (2.97) | 1.6154 (2.02)

7. Secondary Outcome: Montgomery-Asberg Depression Rating Scale
Description: The Montgomery-Åsberg Depression Rating Scale (MADRS) is a psychological questionnaire used by clinicians to assess the severity of depression among patients who have a diagnosis of depression.
  The MADRS depression test includes 10 items and uses a 0 to 6 severity scale. Total score from 0-60. Higher scores indicate increasing depressive symptoms.
Time Frame: baseline and week 14
Population: those who returned for week 14 visit included in data results
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Topiramate | Placebo
Number analyzed (Participants) | 20 | 22
score on a scale
  Baseline | 8.70 (8.29) | 9.54 (6.62)
  week 14: number analyzed (Participants) | 14 | 13
  week 14 | 7.06 (8.54) | 4.69 (5.74)

8. Secondary Outcome: The Hamilton Anxiety Rating Scale
Description: Hamilton Anxiety Rating Scale (HARS) - It consists of 14 items, each defined by a series of symptoms. Each item is rated on a 5-point scale, ranging from 0 (not present) to 4 (severe), with a total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe. Higher score indicates more symptoms.
Time Frame: baseline and week 14
Population: those who returned for week 14 visit included in data results
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Topiramate | Placebo
Number analyzed (Participants) | 20 | 22
score on a scale
  Baseline | 6.35 (3.62) | 7.68 (5.25)
  week 14: number analyzed (Participants) | 14 | 13
  week 14 | 4.94 (5.22) | 5.31 (6.99)

ADVERSE EVENTS:
Arm/Group | Topiramate | Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/22
Other Adverse Events (participants affected / at risk) | 7/20 | 11/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Topiramate (N=20) | Placebo (N=22)
Tiredness (General disorders) | 1 | 2
Headache (General disorders) | 2 | 3
Nausea (Gastrointestinal disorders) | 3 | 4
Shoulder Pain (Musculoskeletal and connective tissue disorders) | 1 | 2

LIMITATIONS AND CAVEATS:
Small sample size and short study duration. Selection bias - sample unrepresentative of PG in the community due to exclusion criteria.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No